CLINICAL TRIAL: NCT05286606
Title: Transforming Older Adult Disability Through Virtual, Peer-Led Community Rehabilitation: Led By MSK Charities
Brief Title: Smart Community Rehabilitation
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Oxford Brookes University (Other)
Collaborators: University of Exeter (Other)
Responsible Party: Principal Investigator, Helen Dawes, Professor, Oxford Brookes University
Other Study IDs: UREC211525
Record Dates: First submitted 2022-02-07; First posted 2022-03-18 (Actual); Last update posted 2022-03-18 (Actual); Status verified 2022-03

CONDITIONS: Musculoskeletal Diseases
MeSH Terms: conditions — Musculoskeletal Diseases | interventions — Exercise; Social Group

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Focus groups: Health Care Professionals (HCP), facilitators, participants in the exercise program will be invited to participate in focus groups to comment on usability/acceptability.
- App users: Users of the exercise program with musculoskeletal conditions have been referred to the exercise program via the charities, all will be participating in a three-month program using the beta version of the app. They will be invited to participate in the program evaluation
  Interventions: Behavioral: Exercise and Social Groups
- Facilitators: Facilitators of the exercise program: The facilitators for the virtual groups have been recruited equally by the charities and are working for GoodBoost to facilitate the exercise program for the app users. They will be invited to participate in the program evaluation

INTERVENTIONS:
Behavioral: Exercise and Social Groups — Participants in the exercise program, which will include a 2-3 time a week 30-45-minute group exercise programme over a 3-month period, 2 x three months. The intervention consists of a 30-45-minute exercise programme. The exercise programme is created by the Good Boost AI based on pre-registration questions or premade sessions, these are either generic sessions with options of strength, aerobic flexibility and balance/coordination exercise with intensity adjusted according to the user's feedback.
  In this program the intervention content is standardised through the Good Boost exercise program. The standard program involves all users to be registered to a single group and to log on to the group, through, zoom, and the facilitator welcomes them. The group then performs the exercise programme they would like to do guided through the app, and afterwards they all meet on a group chat and get peer support.
  Groups: App users

SUMMARY:
Musculoskeletal (MSK) conditions affect 18.8 million people in the UK , accounting for 30% of all GP appointments with combined cost to the NHS of £5bn per year.. It is a highly prevalent and growing umbrella of pain, mobility, function, and inflammatory disorders that account for 40% of all sick leave. Older adults experience almost 2/3rd of MSK prevalence and BAME groups experience high prevalence of certain MSKDs with access inequalities in MSK care and poorer outcomes (Versus Arthritis, 2019). Suffering from a chronic MSK condition is associated with decreased functional capacity, reduction in physical activity and mobility which ultimately results in high costs to health services. In the current climate, the effect of social isolation and redirecting of health care services may prove to expedite the effect of an MSK condition on functional capacity.

There is a large body of evidence for the use of physical activity demonstrates the effectiveness of exercise to treat, manage and prevent MSK conditions . Exercise is one of the primary tools utilised by Physiotherapists throughout the nation and the 'State of Musculoskeletal Health 2019' published by Versus Arthritis cites physical inactivity as a core contributor in growing MSK prevalence and the benefits of exercise for MSK conditions . Access to Physiotherapy services, either due to waiting times, high cost of private care or the non-proximity or remote access to services like Escape Pain are barriers for people living with MSK conditions. Additionally, the primary barrier to anyone living with an MSK condition to being active is pain . As a result, the use of mobile applications to deliver exercise programmes has increased, however, there is a lack of provision for the population of people with MSK problems. Research evidence demonstrates that exercise is highly effective in supporting people living with a joint or pain condition to reduce pain, improve mobility and improve the overall quality of life. However, in the current effect of Covid-19, many people with MSK problems no longer have access to physiotherapy as well as social isolation limiting the opportunities to engage in meaningful physical activity. Trusted by clinicians and patients, MSK charities are the foremost support service to deliver care closer to home, aligning with the NHS strategy.

This project will co-design a solution that is accessible and inclusive by combining cutting-edge technology and MSK charities' networks and expertise, to deliver virtual community MSK rehab, providing an innovative and cost-effective solution to the significant UK and global health challenge. Already overburdened, NHS MSK services are even more pressured due to COVID-19. The project will develop and validate a commercially scalable rehab solution to reduce this pressure. The solution empowers MSK charities to deliver rehab services to beneficiaries through existing, leading-edge AI-powered physiotherapy software. This not only plugs the gap left by long Physiotherapy waiting lists but serves to improve upon existing services by increasing reach and engagement through its community and peer-support aspects. Insight from MSK charities has demonstrated the need for emotional, peer-led and practical rehab solutions that encourage and support patients. The project will be game-changing in driving improved health outcomes for patients and reducing NHS burden and costs.

DETAILED DESCRIPTION:
1.2.1 Background: Musculoskeletal (MSK) conditions affect 18.8 million people in the UK , accounting for 30% of all GP appointments with combined cost to the NHS of £5bn per year. It is a highly prevalent and growing umbrella of pain, mobility, function, and inflammatory disorders that account for 40% of all sick leave. Older adults experience almost 2/3rd of MSK prevalence and BAME groups experience high prevalence of certain MSKDs with access inequalities in MSK care and poorer outcomes (Versus Arthritis, 2019). Suffering from a chronic MSK condition is associated with decreased functional capacity, reduction in physical activity and mobility which ultimately results in high costs to health services. In the current climate, the effect of social isolation and redirecting of health care services may prove to expedite the effect of an MSK condition on functional capacity.

There is a large body of evidence for the use of physical activity demonstrates the effectiveness of exercise to treat, manage and prevent MSK conditions. Exercise is one of the primary tools utilised by Physiotherapists throughout the nation and the 'State of Musculoskeletal Health 2019' published by Versus Arthritis cites physical inactivity as a core contributor in growing MSK prevalence and the benefits of exercise for MSK conditions. Access to Physiotherapy services, either due to waiting times , high cost of private care or the non-proximity or remote access to services like Escape Pain are barriers for people living with MSK conditions. Additionally, the primary barrier to anyone living with an MSK condition to being active is pain. As a result, the use of mobile applications to deliver exercise programmes has increased, however, there is a lack of provision for the population of people with MSK problems. Research evidence demonstrates that exercise is highly effective in supporting people living with a joint or pain condition to reduce pain, improve mobility and improve the overall quality of life. However, in the current effect of Covid-19, many people with MSK problems no longer have access to physiotherapy as well as social isolation limiting the opportunities to engage in meaningful physical activity. Trusted by clinicians and patients, MSK charities are the foremost support service to deliver care closer to home, aligning with the NHS strategy.

This project will co-design a solution that is accessible and inclusive by combining cutting-edge technology and MSK charities' networks and expertise, to deliver virtual community MSK rehab, providing an innovative and cost-effective solution to the significant UK and global health challenge. Already overburdened, NHS MSK services are even more pressured due to COVID-19. The project will develop and validate a commercially scalable rehab solution to reduce this pressure. The solution empowers MSK charities to deliver rehab services to beneficiaries through existing, leading-edge AI-powered physiotherapy software. This not only plugs the gap left by long Physiotherapy waiting lists but serves to improve upon existing services by increasing reach and engagement through its community and peer-support aspects. Insight from MSK charities has demonstrated the need for emotional, peer-led and practical rehab solutions that encourage and support patients. The project will be game-changing in driving improved health outcomes for patients and reducing NHS burden and costs.

1.2.2 Aim: This research project aims to complete product testing, co-production, and research to achieve regulatory approval for public rollout and commercialisation to create a publicly accessible product which will address clinical rehab needs for MSKDs and reduce health inequality. The project will determine the usability, acceptability, and feasibility for use of the developed App.

1.2.3 Objectives: There are two objectives in this study. First one is the usability of the app and second one is the app feasibility

Usability: To discover the barriers and facilitators and potential of using and adopting virtual group digital technology in the management of MSK condition.

Feasibility: to determine the safety, usability and potential benefit of the app

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria app user

Aged over 18

Living with an MSK condition

Is happy to take part in exercise at home

Has not been advised by a health care professional to stop/avoid physical activity and complete the Canadian Physical Activity Questionnaire PARQ

Has an apple (iOS) or Android phone to download the app.

Is happy to take part in the pilot for the duration of the 3-month pilot (if they are signing up for the first quarter (Oct-Jan) or second quarter (Jan-Apr). Over this time that participants will average at least one 30-minute session every two weeks

Is happy to provide feedback on their experience to improve the digital service (through up to 2x virtual focus groups and 2 x online questionnaires)

Is happy to volunteer and consent for their anonymised data to be included in the project research evaluation

2.2.2 Virtual group facilitators (Facilitators)

Sample size (Recruitment phase I; up to n = 10, Recruitment phase III up to 20 depending on requirement based on user recruitment).

Inclusion criteria

These are recruited by the charities, internally and thus inclusion is based on the specific charities

undergone the facilitators training course.

2.2. 3 Focus group

Sample size (Recruitment phase I; up to n = 10. Charities have their own clinical experts and recruitment will from their initially (no advert needed. This group are not study participants but could take part as first app testers to feedback and help in the design) 2.2.2 Virtual group facilitators (Facilitators)

Sample size (Recruitment phase I; up to n = 10, Recruitment phase III up to 20 depending on requirement based on user recruitment).

Inclusion criteria

These are recruited by the charities, internally and thus inclusion is based on the specific charities

undergone the facilitators training course.

2.2. 3 Experts (HCP)

Healthcare professional involved in treatment of MSK condition

Exclusion Criteria:

not meeting the inclusion criteria for each group Under 18 years old Not being familiar with technology

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Users with MSK using the exercise program: In Phase II work package 1: recruitment of the first group of people will be recruited via charities who are collaborating and participating in the Good Boost exercise program, all will participate in a three-month pilot of the beta-app and up to n = 40 of these will be invited to pre and post beta-testing focus groups.
  Facilitators facilitating the program: The facilitators for the virtual groups will be recruited equally by the charities and will work for GoodBoost to facilitate the study for the app users.
  Health Care Professionals (HCP): The focus group will also be recruited at this phase . Ideally initially recruited facilitators and HCPs will complete all phases of the research but additional will be recruited as needed for example in phase III more facilitators possibly will be recruited if user sample size is large. They can be study First testers as a volunteer and will take part in a focus group with two sessions.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2022-02-14 (Actual); Primary Completion 2022-07-14 (Estimated); Study Completion 2022-09-14 (Estimated)

PRIMARY OUTCOMES:
We are performing a program evaluation of the Good Boost exercise program. The primary outcome is measuring the usability of the APP over the program. | 6 months
  We are determining usability as measured by the number of sessions attended.

SECONDARY OUTCOMES:
Health related Quality of life (EQ 5D) | 6 months
  Eq5d
MSK condition musculoskeletal health Questionnaire (MSK-HQ) | 6 month
  MSK condition musculoskeletal health Questionnaire (MSK-HQ)
Physical activity International Physical activity questionnaire.(IPAQ | 6 month
  Physical activity International Physical activity questionnaire.(IPAQ
Functional capacity 2 sit to stand (30 sec) | 6 month
  measured using an IMU sit to stand on the spot
Functional capacity 3 Timed up and go (time) sec ) | 6 month
  measured over a 3 meter course using an IMU
Accessiblity | 6 month
  app usage using interviews and views and opininions
Completion of outcome measures | 6 months
  percentage of completion of the Health related Quality of life (EQ 5D), Physical activity International Physical activity questionnaire.(IPAQ) and MSK condition musculoskeletal health Questionnaire (MSK-HQ).
recrtuitment rate | 6 months
  recruitment rate of the number of people expressing an interest in using the app and registering on the study.
Retention to the research measures | 6 months
  retention as measured by completion outcome measures at follow up

CONTACTS AND LOCATIONS:
Overall Officials: helen Dawes, phd, Principal Investigator — Oxford Brookes University
Locations (1):
- Oxford Brookes, Oxford, United Kingdom

IPD SHARING:
Plan to Share IPD: No